CLINICAL TRIAL: NCT01384955
Title: THE ASSESSMENT OF QUALITY OF LIFE AND FUNCTION OF ADULTS TREATED IN ADOLESCENCE FOR IDIOPATHIC SCOLIOSIS WITH PHYSICAL EXERCISES
Brief Title: HRQoL and Function of Adults Treated in Adolescence for Scoliosis With Physical Exercises
Status: Completed | Type: Observational
Sponsor: Józef Piłsudski University of Physical Education (Other)
Responsible Party: Principal Investigator, Maciej Plaszewski, PhD, Józef Piłsudski University of Physical Education
Other Study IDs: DS.136
Record Dates: First submitted 2011-06-27; First posted 2011-06-29 (Estimated); Last update posted 2015-04-02 (Estimated); Status verified 2015-03

CONDITIONS: Scoliosis
Keywords: scoliosis; physical therapy; long term outcome; pulmonary function; physical fitness; health related quality of life; psychopathology
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- exercise: subjects diagnosed and treated in the Centre of Corrective and Compensatory Gymnastics in Bielsko - Biala, Poland, between 1983 and 1994, with scoliosis - specific exercise program
- control: age and condition - matched subjects, who were diagnosed at the same time, in the same clinic, and by the same physician, and prescribed the same method of physiotherapy, but did not start the exercise treatment

SUMMARY:
We attempt to investigate the influence of physiotherapy and physical activity education applied in adolescence on physical fitness, curve progression, pulmonary function, physical activity and quality of life in adulthood. Quality of life assessment includes mental and social functioning, body image, self - esteem, depression and anxiety surveillance. The follow - up period ranges from 15 to 26 years. Also a group of shorter follow - up of 9 - 13 years is available.

The null hypothesis is that scoliosis specific exercise program applied in adolescence does not influence HRQoL and functioning in adulthood.

DETAILED DESCRIPTION:
Among conservative treatment approaches of adolescent idiopathic scoliosis (AIS), different physiotherapy methods are recommended and popular in some countries (Spain, Germany, Poland), while in others bracing and observation are standard (North America, Australia, the UK, Scandinavia. Neither of the methods have been shown to be definitely effective. Considerable evidence indicates that bracing can lead to psychological stress, poorer body image and self - esteem and reduce overall quality of life in adulthood. As to physiotherapy and physical exercises, such evidence is limited, especially long term follow up studies are not available.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of scoliosis in adolescence
* participation in exercise program in the Centre of Compensatory Gymnastics in Bielsko-Biala in adolescence
* medical records available

Exclusion Criteria:

* contraindications for pulmonary and / or exercise tests
* psychiatric disorders
* recent trauma
* recent traumatic (emotional) event
* contraindications for x-ray exposure

Ages: 22 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Treatment group (retrospection - medical records) - patients diagnosed and / or treated in the Centre of Corrective and Compensatory Gymnastics in Bielsko - Biala, Poland, between 1983 and 1994. Diagnosis: idiopathic scoliosis (IS) - adolescent idiopathic scoliosis (AIS) or early onset idiopathic scoliosis (EOIS) A comparison (control) group: patients with IS, age - and condition - matched, who were diagnosed at the same time, in the same clinic, and by the same physician, and prescribed the same method of physiotherapy, but did not start the exercise treatment.
Sampling Method: Non-Probability Sample
Enrollment: 143 (Actual)
Dates: Start 2010-01; Primary Completion 2013-04 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
health related quality of life | one time point
  generic and condition-specific questionnaires

SECONDARY OUTCOMES:
pulmonary function | one time point
  spirometry, total lung capacity
physical fitness | one time point
  cycloergometric submaximal physical working capacity test
curve progression | two time points: data from medical records (past) and present meausserements
  x-ray, Cobb angle, trunk rotation, scoliometer

OTHER OUTCOMES:
psychopathology | one time point
  questionnaires / inventories of mental heath (e.g. depression, anxiety)

CONTACTS AND LOCATIONS:
Overall Officials: Maciej Plaszewski, PhD, Study Director — Faculty of Physical Education and Sport in Biala Podlaska, University School of Physical Education, Warsaw, Poland
Locations (1):
- Faculty of Physiotherapy, WSA, Bielsko-Biala, Poland

REFERENCES:
- [Derived] Plaszewski M, Cieslinski I, Kowalski P, Truszczynska A, Nowobilski R. Does scoliosis-specific exercise treatment in adolescence alter adult quality of life? ScientificWorldJournal. 2014;2014:539671. doi: 10.1155/2014/539671. Epub 2014 Nov 10. PMID 25436225
- [Derived] Plaszewski M, Cieslinski I, Nowobilski R, Kotwicki T, Terech J, Furgal M. Mental health of adults treated in adolescence with scoliosis-specific exercise program or observed for idiopathic scoliosis. ScientificWorldJournal. 2014 Jan 20;2014:932827. doi: 10.1155/2014/932827. eCollection 2014. PMID 24574935